CLINICAL TRIAL: NCT06698913
Title: Feasibility and Efficacy of Automated Lateral Decubitus Therapy in Hypoxemic Respiratory Failure
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 44692221.5.0000.0068
Record Dates: First submitted 2024-10-23; First posted 2024-11-21 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-09

CONDITIONS: Respiratory Insufficiency; ARDS; Post Cardiac Surgery Patients; Hypoxemic Respiratory Failure
Keywords: alveolar recruitment; post cardiac surgery; lateral position; Hypoxemic Respiratory Failure
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Intervention Model Description: In Sample 1, intervention group patients had ventilator settings adjusted with PEEP based on BMI, followed by a 2 cmH2O increase and 20 minutes in a lateral position at 30 degrees for lung recruitment, monitored by plethysmogram. PEEP was increased up to 4 cmH2O as needed. Afterward, patients returned to supine, and the process was repeated on the other side. The control group had similar ventilator settings but stayed supine. Both groups had an alveolar recruitment maneuver with increased pressures. In Sample 2, all patients underwent a 2-minute recruitment maneuver, followed by a 5-minute PEEP titration. The EIT-PEEP was identified and selected as the first PEEP above the crossing point of collapse and hyperdistension curves. Patients were then randomized, and PEEP was increased progressively based on randomization. The intervention group avoided traditional recruitment maneuvers, increasing PEEP gradually. This was followed by 4 hours of observation and a 24-hour follow-up
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Lateral Positioning (Experimental): Sample1- Ventilator settings where adjusted with PEEP based on BMI, followed by a 2 cmH2O increase and 20 minutes in a lateral position at 30 degrees for lung recruitment for both sides. And at the end were subjected to an alveolar recruitment maneuver with pressure increases up to a plateau pressure of 45 cmH2O. Sample2- A recruitment maneuver followed by PEEP titration is performed, selecting the PEEP that is above the crossing point between the collapse and hyperdistension curves provided by EIT. And the the PEEP-ARDSNet will be selected according to the low PEEP-FIO2 table from the ARDSNet protocol. Observations are made at 4 and 24 hours, with PEEP at 24 hours adjusted to the level identified by EIT.
  Interventions: Procedure: Rotational Therapy
- Control Group (No Intervention): Sample 1- The ventilator settings adjusted with PEEP based on BMI and remained in the supine position for the entire time. And at the end were subjected to an alveolar recruitment maneuver with pressure increases up to a plateau pressure of 45 cmH2O.Sample 2- A recruitment maneuver followed by PEEP titration is performed, selecting the PEEP that is above the crossing point between the collapse and hyperdistension curves provided by EIT. And the the PEEP-ARDSNet will be selected according to the low PEEP-FIO2 table from the ARDSNet protocol. Observations are made at 4 and 24 hours, with PEEP at 24 hours adjusted to the level identified by EIT

INTERVENTIONS:
Procedure: Rotational Therapy — Sample1- Ventilator settings where adjusted with PEEP based on BMI, followed by a 2 cmH2O increase and 20 minutes in a lateral position at 30 degrees for lung recruitment for both sides. And at the end were subjected to an alveolar recruitment maneuver with pressure increases up to a plateau pressure of 45 cmH2O. Sample2- A recruitment maneuver followed by PEEP titration is performed, selecting the PEEP that is above the crossing point between the collapse and hyperdistension curves provided by EIT. And the the PEEP-ARDSNet will be selected according to the low PEEP-FIO2 table from the ARDSNet protocol. Observations are made at 4 and 24 hours, with PEEP at 24 hours adjusted to the level identified by EIT.
  Arms: Lateral Positioning

SUMMARY:
The mortality of patients with acute respiratory distress syndrome (ARDS) remains high despite recent advances in lung-protective strategies and even after the overall improvement in intensive care (management of sepsis, hemodynamics, organ failure, and control of nosocomial infections). The use of mechanical ventilation (MV) plays a fundamental therapeutic role in this scenario. It allows for respiratory muscle rest, maintenance of oxygen transport to tissues, elimination of CO2 production, and finally, lung rest and protection in patients with excessive ventilatory demand.

On the other hand, recent studies have also shown that MV can cause iatrogenic injury and inflammation in the lung parenchyma, imposing a significant mechanical energy load and dissipation in the lung parenchyma (mechanotransduction). This effect is more pronounced in patients with low lung compliance or in those receiving inadvertently high tidal volumes, resulting in high distending pressure. Thus, despite being life-saving in the short term, MV may perpetuate or exacerbate pre-existing lung injury.

Various strategies have been proposed to aid in the ventilatory management of patients with ARDS. Among them, the use of higher PEEP values and the prone position have proven beneficial, especially when resulting in the stabilization of diseased alveoli or even promoting the recruitment of new alveolar units, associated with improved gas exchange. Both maneuvers, however, involve considerable risks: PEEP often causes impairments to venous return, and the prone position presents technical/logistical limitations for its widespread use, or even severe adverse effects during its implementation (ocular injury, accidental extubation, arrhythmias, catheter disconnection, etc.).

The hypothesis of this study is that automated lateral decubitus positioning (performed by a rotational bed with proper patient support), guided by monitoring through Electrical Impedance Tomography (EIT), could replace or minimize the need for prone positioning or the need for higher PEEPs in critical patients, resulting in effective alveolar recruitment and improvements in gas exchange, compliance, and lung aeration without affecting the hemodynamic condition.

DETAILED DESCRIPTION:
The objective will be to estimate the efficacy and validate the feasibility of this alveolar recruitment protocol through the automated rotation of the patient, without the need for high airway pressures.Also the aim to demonstrate that this protocol is safe, with fewer repercussions on the hemodynamics of critically ill patients. To achieve this, a prospective, randomized study were conduct in two populations of critically ill patients: Sample-1) patients in the postoperative period of cardiac surgery, with a PF ratio of less than 250 (N=50 patients) admitted to the post-anesthesia care unit of Incor for extubation, and Sample-2) patients with ARDS or acute hypoxemic respiratory failure, with a PF ratio of less than 250, requiring mechanical ventilation (N=30 additional patients), and necessarily presenting an asymmetric (>65%/35%) distribution of ventilation on the functional map of Electrical Impedance Tomography (EIT) while in the supine position. A stratified randomization (1:1) within each of these samples of 30 patients will be done by computer.

For Sample 1 - the control group will undergo an ARDSNet-type ventilatory strategy, with PEEP adjustment according to BMI, based on previous studies that evaluated PEEP titrated by EIT in relation to BMI; and for Sample 2 - the ARDSNet-type ventilatory strategy, with PEEP adjustment according to the "low PEEP/FIO2" oxygenation table. All patients will remain on mechanical ventilation for at least 4 hours and will be monitored with EIT throughout the study. In postoperative patients, the rotation of the treatment group will follow the sequence "supine - lateral - supine - lateral - supine," with 10 minutes in each supine position and 20 minutes in each lateral position, and the first rotated side is defined as the lung with less ventilation being placed in a non-dependent position with a maximum PEEP of 24 cmH2O. In patients with asymmetric injury (acute hypoxemic respiratory failure), the lateralization sequence will be "supine-lateral with the better lung dependent-supine," meaning that the rotation will be unilateral, with 20-minute lateral position times alternated with another 10 minutes in the supine position. Recruitment maneuvers routinely used by the institution may be used as a rescue for any patient and will be mandatory at the end of the 4-hour study period in all postoperative patients (Sample 1, both treatment arms). The maneuvers will be performed with controlled pressure ventilation, a maximum PEEP of 30 cmH2O, with maximum inspiratory pressures of 50 cmH2O, for a maximum time of 30 seconds. These maneuvers will not be applied to patients with asymmetric injury (Sample 2, acute hypoxemic respiratory failure).

The main variables for comparison between the arms of each population sample will be: a) lung collapse and hyperdistension, b) shunt and PF ratio, c) ventilatory ratio (as a "surrogate" for dead space), d) global lung mechanics, e) regional mechanics by EIT, and f) continuous measurements of cardiac output (Volume-View, Baxter), frequency, and mean arterial pressure. These variables will be collected during the baseline period and after the recruitment maneuver for Sample 1, and after 24 hours of intervention for Sample 2.

The main hypothesis is that rotational therapy can increase regional transpulmonary pressure (in the non-dependent region after rotation), resulting in effective alveolar recruitment, evidenced by an improvement in PF ratio, global compliance, and regional compliance after returning to the supine position in both patient populations. In the case of patients with asymmetric lung injury (Sample 2), a effect is expecting within the following 24 hours compared to the control therapy. In the case of patients with symmetric injury, these effects can also be compared with the effects obtained by the more aggressive and traditional recruitment maneuver to be performed at the end of the observation period. As a secondary hypothesis, it was to intend to demonstrate that the therapy will cause minimal hemodynamic impairment compared to the control arm, and also less hemodynamic impairment when compared to the traditional recruitment maneuver at the end of the study (for postoperative patients).

ELIGIBILITY:
Inclusion Criteria:

Sample 1-

* Patients under mechanical ventilation
* Immediate postoperative period of open-heart valve surgery and myocardial revascularization
* PaO2/FiO2 ratio ≤ 250 mmHg (calculated from values obtained in arterial blood gas analysis)
* Values collected with:

FiO2 ≥ 0.6 PEEP ≥ 8 cmH2O

Sample 2 -

* Patients under controlled/assisted mechanical ventilation, not yet eligible for weaning
* PaO2/FiO2 ratio < 250 mmHg (calculated using arterial blood gas values)
* Values collected with:

FiO2 = 0.6 PEEP > 5 cmH2O

* Acute condition onset less than 2 weeks ago
* Mechanical ventilation duration of less than 1 week
* Asymmetric ventilation distribution (65%/35%) on the functional map from Electrical Impedance Tomography (EIT) in the supine position

Both Samples:

Exclusion Criteria:

* Need for norepinephrine ≥ 1 mcg/kg/min or mean arterial pressure ≤ 65 mmHg;
* Cardiac arrhythmias or bleeding leading to hemodynamic instability;
* Need for surgical revision and/or mechanical circulatory assistance;
* Contraindication to hypercapnia, such as intracranial hypertension or acute coronary syndrome;
* Neurological diseases or symptoms, such as a history of seizures;
* Dependence on a cardiac pacemaker;
* Air leakage through chest drains, undrained pneumothorax, or subcutaneous emphysema;
* Previous lung disease or surgery, or use of home oxygen therapy;
* Comorbidities with a life expectancy < 6 months;
* Pulmonary artery systolic pressure > 45 mmHg;
* Myocardial revascularization using the mammary artery;
* Medical refusal for the patient's participation in the study.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2021-12-13 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Lung Collapse | Right before first lateralization, 10 minutes after the first lateralization, 10 minutes after the second lateralization, 10 minutes after the alveolar recruitment maneuver using the increase of pressures.
  Lung Collapse will be measured using the information provided by the EIT that uses the Costa method
Lung compliance | Right before first lateralization, 10 minutes after the first lateralization, 10 minutes after the second lateralization, 10 minutes after the alveolar recruitment maneuver using the increase of pressures.
  Lung compliance (mL/cmH2O) will be measured using the information provided by the EIT that uses the movement equation
Oxygenation | Right before first lateralization, 10 minutes after the first lateralization, 10 minutes after the second lateralization, 10 minutes after the alveolar recruitment maneuver using the increase of pressures.
  Oxigenation will be assessed using the partial pressure arterial oxygen/fraction inspired oxygen ratio. Partial pressure arterial oxygen measured in the blood sample at the of each step and the fraction inspired oxygen set during the blood sample collection will be used.
Shunt | Right before first lateralization, 10 minutes after the first lateralization, 10 minutes after the second lateralization, 10 minutes after the alveolar recruitment maneuver using the increase of pressures.
  Oxygenation will be assessed using the partial pressure arterial oxygen/fraction inspired oxygen at 1 ratio and partial pressure arterial oxygen and partial pressure of oxygen in venous blood will be collected an calculated manual using the formula Q/Qt= (CcO2-Ca02)-(CcO1-CvO2) where CcO2 (Pulmonary end-capillary O2 content); CvO2 (Mixed venous O2 content); CaO2(Arterial O2 content).
Driving Pressure | Right before first lateralization, 10 minutes after the first lateralization, 10 minutes after the second lateralization, 10 minutes after the alveolar recruitment maneuver using the increase of pressures.
  Driving Pressure (cmH2O) will be measured using the information provided by the EIT that uses the movement equation
End Expiratory Lung Volume | Right before first lateralization, 10 minutes after the first lateralization, 10 minutes after the second lateralization, 10 minutes after the alveolar recruitment maneuver using the increase of pressures.
  will be measured using the information provided by the Electrical Tomography Impedance
Lung Hyperextension | Right before first lateralization, 10 minutes after the first lateralization, 10 minutes after the second lateralization, 10 minutes after the alveolar recruitment maneuver using the increase of pressures.
  Lung Hyperextension (%) will be measured using the information provided by the EIT that uses the Costa method
Plateau Pressure | Right before first lateralization, 10 minutes after the first lateralization, 10 minutes after the second lateralization, 10 minutes after the alveolar recruitment maneuver using the increase of pressures.
  Plateau Pressure( cmH2O) will be measured using the information provided by the EIT that uses the movement equation
Ventilatory Distribution | Right before first lateralization, 10 minutes after the first lateralization, 10 minutes after the second lateralization, 10 minutes after the alveolar recruitment maneuver using the increase of pressures.
  will be measured using the information provided by the Electrical Tomography Impedance

SECONDARY OUTCOMES:
Stroke Volume | the specific time was in each supine position, three at total; during the recruitment maneuver; after 5 and 15 minutes after both lateralization and the record throughout the duration of the protocol in the 20seconds of period of time
  The hemodynamics were assessed through Stroke Volume using the EV1000™ clinical monitoring platform.
Diastolic Blood Pressure | the specific time was in each supine position, three at total; during the recruitment maneuver; after 5 and 15 minutes after both lateralization and
  The hemodynamics were assessed through Diastolic Blood Pressure using the multiparameter monitor DX-2020 (Dixtal, São Paulo, Brazil).
Stroke Volume Index | the specific time was in each supine position, three at total; during the recruitment maneuver; after 5 and 15 minutes after both lateralization and the record throughout the duration of the protocol in the 20seconds of period of time
  The hemodynamics were assessed through Stroke Volume Index using the EV1000™ clinical monitoring platform.
Cardiac Index | the specific time was in each supine position, three at total; during the recruitment maneuver; after 5 and 15 minutes after both lateralization and the record throughout the duration of the protocol in the 20seconds of period of time
  The hemodynamics were assessed through Cardiac Index using the EV1000™ clinical monitoring platform.
Cardiac Output | the specific time was in each supine position, three at total; during the recruitment maneuver; after 5 and 15 minutes after both lateralization and the record throughout the duration of the protocol in the 20seconds of period of time
  The hemodynamics were assessed through Cardiac Output using the EV1000™ clinical monitoring platform.
Systolic Volume Variation | the specific time was in each supine position, three at total; during the recruitment maneuver; after 5 and 15 minutes after both lateralization and the record throughout the duration of the protocol in the 20seconds of period of time
  The hemodynamics were assessed through Systolic Volume Variation using the EV1000™ clinical monitoring platform.
Mean Arterial Pressure | the specific time was in each supine position, three at total; during the recruitment maneuver; after 5 and 15 minutes after both lateralization and the record throughout the duration of the protocol in the 20seconds of period of time
  The hemodynamics were assessed through Mean Artial Pressure using the EV1000™ clinical monitoring platform for continous record and the the multiparameter monitor DX-2020 (Dixtal, São Paulo, Brazil) for especifics times of colleted data.
Pulse Rate | the record throughout the duration of the protocol in the 20seconds of period of time
  The hemodynamics were assessed through Pulse Rate using the EV1000™ clinical monitoring platform.
Systolic Blood Pressure | the specific time was in each supine position, three at total; during the recruitment maneuver; after 5 and 15 minutes after both lateralization and
  The hemodynamics were assessed through Diastolic Blood Pressure using the multiparameter monitor DX-2020 (Dixtal, São Paulo, Brazil).
Heart Rate | the specific time was in each supine position, three at total; during the recruitment maneuver; after 5 and 15 minutes after both lateralization.
  The hemodynamics were assessed through Diastolic Blood Pressure using the multiparameter monitor DX-2020 (Dixtal, São Paulo, Brazil).

CONTACTS AND LOCATIONS:
Overall Officials: Marcelo BP, MD PhD, Principal Investigator — University of Sao Paulo General Hospital
Locations (1):
- Instituto do Coração do Hospital das Clínicas da Faculdade de Medicina da USP, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pereira SM, Tucci MR, Morais CCA, Simoes CM, Tonelotto BFF, Pompeo MS, Kay FU, Pelosi P, Vieira JE, Amato MBP. Individual Positive End-expiratory Pressure Settings Optimize Intraoperative Mechanical Ventilation and Reduce Postoperative Atelectasis. Anesthesiology. 2018 Dec;129(6):1070-1081. doi: 10.1097/ALN.0000000000002435. PMID 30260897
- [Background] Costa EL, Lima RG, Amato MB. Electrical impedance tomography. Curr Opin Crit Care. 2009 Feb;15(1):18-24. doi: 10.1097/mcc.0b013e3283220e8c. PMID 19186406
- [Background] Hewitt N, Bucknall T, Faraone NM. Lateral positioning for critically ill adult patients. Cochrane Database Syst Rev. 2016 May 12;2016(5):CD007205. doi: 10.1002/14651858.CD007205.pub2. PMID 27169365
- [Background] Tongyoo S, Vilaichone W, Ratanarat R, Permpikul C. The effect of lateral position on oxygenation in ARDS patients: a pilot study. J Med Assoc Thai. 2006 Nov;89 Suppl 5:S55-61. PMID 17718246
- [Background] Remolina C, Khan AU, Santiago TV, Edelman NH. Positional hypoxemia in unilateral lung disease. N Engl J Med. 1981 Feb 26;304(9):523-5. doi: 10.1056/NEJM198102263040906. No abstract available. PMID 6779161
- [Background] Scholten EL, Beitler JR, Prisk GK, Malhotra A. Treatment of ARDS With Prone Positioning. Chest. 2017 Jan;151(1):215-224. doi: 10.1016/j.chest.2016.06.032. Epub 2016 Jul 8. PMID 27400909
- [Background] Fessler HE, Talmor DS. Should prone positioning be routinely used for lung protection during mechanical ventilation? Respir Care. 2010 Jan;55(1):88-99. PMID 20040127
- [Background] Puybasset L, Cluzel P, Chao N, Slutsky AS, Coriat P, Rouby JJ. A computed tomography scan assessment of regional lung volume in acute lung injury. The CT Scan ARDS Study Group. Am J Respir Crit Care Med. 1998 Nov;158(5 Pt 1):1644-55. doi: 10.1164/ajrccm.158.5.9802003. PMID 9817720
- [Background] Pelosi P, D'Andrea L, Vitale G, Pesenti A, Gattinoni L. Vertical gradient of regional lung inflation in adult respiratory distress syndrome. Am J Respir Crit Care Med. 1994 Jan;149(1):8-13. doi: 10.1164/ajrccm.149.1.8111603.
- [Background] Malbouisson LM, Busch CJ, Puybasset L, Lu Q, Cluzel P, Rouby JJ. Role of the heart in the loss of aeration characterizing lower lobes in acute respiratory distress syndrome. CT Scan ARDS Study Group. Am J Respir Crit Care Med. 2000 Jun;161(6):2005-12. doi: 10.1164/ajrccm.161.6.9907067. PMID 10852781
- [Background] Lai-Fook SJ, Rodarte JR. Pleural pressure distribution and its relationship to lung volume and interstitial pressure. J Appl Physiol (1985). 1991 Mar;70(3):967-78. doi: 10.1152/jappl.1991.70.3.967. PMID 2033012
- [Background] Writing Group for the Alveolar Recruitment for Acute Respiratory Distress Syndrome Trial (ART) Investigators; Cavalcanti AB, Suzumura EA, Laranjeira LN, Paisani DM, Damiani LP, Guimaraes HP, Romano ER, Regenga MM, Taniguchi LNT, Teixeira C, Pinheiro de Oliveira R, Machado FR, Diaz-Quijano FA, Filho MSA, Maia IS, Caser EB, Filho WO, Borges MC, Martins PA, Matsui M, Ospina-Tascon GA, Giancursi TS, Giraldo-Ramirez ND, Vieira SRR, Assef MDGPL, Hasan MS, Szczeklik W, Rios F, Amato MBP, Berwanger O, Ribeiro de Carvalho CR. Effect of Lung Recruitment and Titrated Positive End-Expiratory Pressure (PEEP) vs Low PEEP on Mortality in Patients With Acute Respiratory Distress Syndrome: A Randomized Clinical Trial. JAMA. 2017 Oct 10;318(14):1335-1345. doi: 10.1001/jama.2017.14171. PMID 28973363
- [Background] Meade MO, Cook DJ, Guyatt GH, Slutsky AS, Arabi YM, Cooper DJ, Davies AR, Hand LE, Zhou Q, Thabane L, Austin P, Lapinsky S, Baxter A, Russell J, Skrobik Y, Ronco JJ, Stewart TE; Lung Open Ventilation Study Investigators. Ventilation strategy using low tidal volumes, recruitment maneuvers, and high positive end-expiratory pressure for acute lung injury and acute respiratory distress syndrome: a randomized controlled trial. JAMA. 2008 Feb 13;299(6):637-45. doi: 10.1001/jama.299.6.637. PMID 18270352
- [Background] Terragni PP, Rosboch G, Tealdi A, Corno E, Menaldo E, Davini O, Gandini G, Herrmann P, Mascia L, Quintel M, Slutsky AS, Gattinoni L, Ranieri VM. Tidal hyperinflation during low tidal volume ventilation in acute respiratory distress syndrome. Am J Respir Crit Care Med. 2007 Jan 15;175(2):160-6. doi: 10.1164/rccm.200607-915OC. Epub 2006 Oct 12. PMID 17038660
- [Background] Slutsky AS, Ranieri VM. Ventilator-induced lung injury. N Engl J Med. 2013 Nov 28;369(22):2126-36. doi: 10.1056/NEJMra1208707. No abstract available. PMID 24283226
- [Background] Amato MB, Barbas CS, Medeiros DM, Magaldi RB, Schettino GP, Lorenzi-Filho G, Kairalla RA, Deheinzelin D, Munoz C, Oliveira R, Takagaki TY, Carvalho CR. Effect of a protective-ventilation strategy on mortality in the acute respiratory distress syndrome. N Engl J Med. 1998 Feb 5;338(6):347-54. doi: 10.1056/NEJM199802053380602. PMID 9449727
- [Background] Acute Respiratory Distress Syndrome Network; Brower RG, Matthay MA, Morris A, Schoenfeld D, Thompson BT, Wheeler A. Ventilation with lower tidal volumes as compared with traditional tidal volumes for acute lung injury and the acute respiratory distress syndrome. N Engl J Med. 2000 May 4;342(18):1301-8. doi: 10.1056/NEJM200005043421801. PMID 10793162
- [Background] ARDS Definition Task Force; Ranieri VM, Rubenfeld GD, Thompson BT, Ferguson ND, Caldwell E, Fan E, Camporota L, Slutsky AS. Acute respiratory distress syndrome: the Berlin Definition. JAMA. 2012 Jun 20;307(23):2526-33. doi: 10.1001/jama.2012.5669. PMID 22797452
- [Background] Costa EL, Amato MB. The new definition for acute lung injury and acute respiratory distress syndrome: is there room for improvement? Curr Opin Crit Care. 2013 Feb;19(1):16-23. doi: 10.1097/MCC.0b013e32835c50b1. PMID 23235543
- [Background] Matthay MA, Zemans RL, Zimmerman GA, Arabi YM, Beitler JR, Mercat A, Herridge M, Randolph AG, Calfee CS. Acute respiratory distress syndrome. Nat Rev Dis Primers. 2019 Mar 14;5(1):18. doi: 10.1038/s41572-019-0069-0. PMID 30872586